CLINICAL TRIAL: NCT00670410
Title: A Pilot Study of Sequential Autologous Stem Cell Transplantation and Immunotherapy With Reduced Intensity Allogeneic Stem Cell Transplant for High Risk Neuroblastoma
Brief Title: Autologous Transplant Followed by Allogeneic Transplant for High Risk Neuroblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAA7937; CHNY-01-502 (Other: CUMC)
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Autologous Transplant; Allogeneic Transplant; Immunotherapy
MeSH Terms: conditions — Neuroblastoma | interventions — Busulfan; thymoglobulin; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - Related Donor (Experimental): Related donor transplant: Patients with a related donor (5/6 or 6/6 HLA matched) will receive immunotherapy with a non-myeloablative preparative regimen of Busulfan and Fludarabine followed by allogeneic stem cell transplant (AlloSCT).
  Interventions: Procedure: Related donor transplant; Drug: Busulfan; Drug: Fludarabine
- Arm B - Cord Blood Donor (Experimental): Unrelated cord blood transplant: Patients without a related donor will receive immunotherapy with a non-myeloablative preparative regimen of busulfan and fludarabine followed by allogeneic stem cell transplant (AlloSCT) with either an unrelated umbilical cord blood donor (4/6, 5/6, or 6/6 HLA matched), or a related umbilical cord blood donor (3/6, 4/6, 5/6, or 6/6 HLA matched). Patients will receive Thymoglobulin ((rabbit) Anti-Thymocyte Globulin (ATG)) during the preparative regimen. GVHD prophylaxis will be Tacrolimus and mycophenolate mofetil (MMF).
  Interventions: Procedure: Cord blood transplant; Drug: Busulfan; Drug: Thymoglobulin; Drug: Fludarabine

INTERVENTIONS:
Procedure: Related donor transplant — Patients with a related donor will get reduced intensity transplant conditioning with busulfan and fludarabine.
  Arms: Arm A - Related Donor
Procedure: Cord blood transplant — Patients with a matched cord blood donor will get reduced intensity conditioning with busulfan, fludarabine, and ATG.
  Arms: Arm B - Cord Blood Donor
Drug: Busulfan — Busulfan (Busulfex) [4mg/kg/dose for patients < 4 years; 3.2 mg/kg/dose for patients > 4 years] will be given IV in 0.9% sodium chloride or D5W to a final concentration > 0.5 mg/mL solution for infusion equal to 10 times the volume of diluent to Busulfex, through a central venous access device over 3 hours once daily.
  Other Names: Busulfex®
Drug: Thymoglobulin — Patients with an umbilical cord blood donor will also receive Thymoglobulin (ATG-rabbit) during the preparative regimen.
  Other Names: ATG-rabbit
  Arms: Arm B - Cord Blood Donor
Drug: Fludarabine — Fludarabine 30 mg/m2 x 5 days, total dose = 150 mg/m2. Patients < 12 kg will receive Fludarabine 1 mg/kg x 5 days, total dose = 5 mg/kg. Fludarabine will be given IV in 100 ml (or to a concentration of 1 mg/mL) of D5W or 0.9% sodium chloride, and infused over 30 min on Days -6 to 2.
  Other Names: Fludara®

SUMMARY:
Neuroblastoma is a malignant tumor of the sympathetic nervous system. It is the second most common malignant tumor of childhood. Although modest advances have been made over the past 20 years children with high-risk neuroblastoma continue to have an unsatisfactory long-term survival. This study will administer induction chemotherapy followed by high-dose (myeloablative) chemotherapy with autologous stem cell transplantation, followed by radiation therapy, then immunotherapy with a non myeloablative allogeneic stem cell transplant for treatment of neuroblastoma. The purpose of this clinical research trial is to study the feasibility of giving immunotherapy with a non-myeloablative allogeneic transplant (NAT/AlloSCT), following myeloablative therapy and autologous stem cell transplant (MAT/AutoSCT). This study will also determine the side effects as well as the response rate for each group of patients (treatment arm).

DETAILED DESCRIPTION:
Despite the modest advances made over the past two decades with the addition of more intensive chemotherapy and high dose myeloablative therapy with allogeneic or autologous bone marrow transplantation, children with high-risk neuroblastoma continue to have an unsatisfactory long-term survival. The current survival for a child > 1 year of age at diagnosis with stage 4 neuroblastoma is only 20-35% 1,7. The overall treatment plan for high-risk patients with neuroblastoma will be:

Induction Therapy Intensive induction chemotherapy with the cardioprotectant dexrazoxane (Zinecard), vincristine, doxorubicin (Adriamycin), and cyclophosphamide (ZVAC), alternating with cisplatin and etoposide (CiE). Patients who receive induction chemotherapy on an alternate protocol and achieve a CR, VGPR, or PR will also be eligible for entry to receive consolidation therapy and AlloSCT immunotherapy after discussion and approval of the Principal Investigators ).

Consolidation Therapy with AutoSCT Consolidation therapy with a myeloablative preparative regimen of carboplatin, thiotepa, and topotecan (CaTT) followed by AutoSCT with PBSCs (CD34+ selection optional).

Immunotherapy with Non-myeloablative AlloSCT Immunotherapy with a non-myeloablative preparative regimen of busulfan and fludarabine followed by AlloSCT with either: (Arm A) a related donor (5/6 or 6/6 HLA matched); or (Arm B) an umbilical cord blood donor (unrelated 4/6, 5/6, or 6/6 HLA matched, or related 3/6, 4/6, 5/6, or 6/6 HLA matched). Patients with an umbilical cord blood donor will also receive Thymoglobulin (ATG-rabbit) during the preparative regimen. GVHD prophylaxis will consist of Tacrolimus and mycophenolate mofetil (MMF).

Maintenance Therapy Patients with a related donor who have persistent disease detected prior to NAT/AlloSCT will be assigned to Arm A1 and will receive two courses of DLI, followed by cis-RA for 6 cycles. Patients with a related donor with no persistent disease detected prior to NAT/AlloSCT will be assigned to Arm A2 and receive cis-RA for 6 cycles. Patients with an umbilical cord blood donor will receive cis-RA for 6 cycles.

Radiation Therapy Due to the potential risk of increased GVHD following radiation therapy, local radiation therapy to the primary tumor site (21 Gy) and metastatic sites, will be given after NAT/AlloSCT for patients on Arm A2 and Arm B, and prior to cis-RA therapy. Radiation therapy will be given following DLI in Arm A1, and prior to cis-RA therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age be < 30 years of age at the time of initial diagnosis.
* Patients must have a diagnosis of neuroblastoma (ICD-O morphology 9500/3) verified by histology and/or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites. Patients with the following disease stages at diagnosis are eligible, if they meet the other specified criteria. The revised International Neuroblastoma Staging System (INSS) will be used to stage all patients 58. (See 14.3 for risk assignment).
* Patients with newly diagnosed neuroblastoma and age > 547 days with the following:

  * INSS Stage 4 neuroblastoma regardless of biologic factors
  * INSS Stage 2A/2B with MYCN amplification (> 10)
  * INSS Stage 3 with MYCN amplification (> 10) OR Unfavorable histology
* Patients with newly diagnosed neuroblastoma and age < 365 days with the following:

  * INSS Stage 3, 4, OR 4S neuroblastoma AND MYCN amplification (> 10).
* Patients with newly diagnosed Neuroblastoma and age 365 - <547 days with the following:

  * INSS Stage 3 with MYCN amplification (> 10)
  * INSS Stage 4 with MYCN amplification (> 10) OR with deoxyribonucleic acid (DNA) Index (ploidy) = 1 OR with Unfavorable histology
* Patients > 365 days with INSS Stage 1, 2, and 4S who have progressed to Stage 4.
* Newly Diagnosed patients should be entered on this study within 4 weeks of diagnosis, or after receiving only one cycle of intermediate dose chemotherapy for patients initially treated on/according to the low or intermediate risk Children's Oncology Group (COG) neuroblastoma studies, or within 4 weeks of progression to Stage 4 for INSS Stage 1, 2, 4S.
* Patients treated with alternative induction regimens and/or consolidation regimens (AutoSCT) who were not enrolled at diagnosis but who achieve a complete response (CR), very good partial response (VGPR), partial response (PR), or minimal response (MR) and meet all other criteria will be eligible for either the consolidation MAT/AutoSCT and NAT/AlloSCT immunotherapy or NAT/AlloSCT, which ever is clinically appropriate after discussion with the Principal Investigators.
* Liver Function: alanine aminotransferase (ALT) and bilirubin < 3x normal
* Cardiac Function: Shortening fraction > 27%, or ejection fraction > 47%, no clinical congestive heart failure.
* Renal Function: Creatinine clearance and/or glomerular filtration rate (GFR) > 60 ml/min/1.73m2.
* Hematologic Function: Patients must have adequate hematopoietic function (absolute neutrophil count (ANC) > 1000/mm3 and platelets > 100,000/mm3) unless inadequate hematopoiesis documented to be due to bone marrow involvement with tumor (> 10% tumor infiltration).

Exclusion Criteria:

* Patients who are pregnant. Patients of childbearing potential must practice an effective method of birth control while participating on this study.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2003-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Rate of engraftment following NAT/AlloSCT from either a related donor or umbilical cord donor. | 1 year
  The distribution of the time to neutrophil and platelet engraftment following consolidation (myeloablative) and intensification (non-ablation) will be estimated using the product-limit method of the Kaplan and Meier.
Progression Free Survival (PFS) in patients with high-risk neuroblastoma receiving sequential MAT/AutoSCT and NAT/AlloSCT. | 5 years
  Progression Free (PFS) will be estimated using the product limit method of Kaplan and Meier.
Overall Survival (OS) in patient with high-risk neuroblastoma receiving sequential MAT/AutoSCT and NAT/AlloSCT. | 5 years
  Overall Survival (OS) will be estimated using the product limit method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Darrell Yamashiro, MD, Study Chair — Columbia University
Locations (1):
- Columbia Presbyterian Medical Center, Morgan Stanley Children's Hospital New York Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Unknown.